CLINICAL TRIAL: NCT03617835
Title: Relative Bioavailability, Safety, and Tolerability Following Subcutaneous Injection of Different Doses of BI 655130 and Different Injection Sites in Healthy Male and Female Subjects (a Single Dose, Mono-centric, Open-label Study in Matched-group Design).
Brief Title: A Study in Healthy People to Measure the Amount of BI 655130 in the Blood After Injecting Different Doses Into Different Parts of the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0029; 2018-001074-18 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R - Low dose of BI 655130 Periumbilical (Experimental): Single low dose of BI 655130 administered as one single subcutaneous injection (given as 1 x 2 milliliter (mL)) in the periumbilical region following an overnight fast of at least 10 hours.
  Interventions: Drug: R - Low dose of BI 655130
- T1 - Low dose of BI 655130 Periumbilical (left and right) (Experimental): Single low dose of BI 655130 administered as two single subcutaneous injections (given as 2 x 1 milliliter (mL)) in the periumbilical region (left and right) following an overnight fast of at least 10 hours.
  Interventions: Drug: T1 - Low dose of BI 655130
- T2 - Low dose of BI 655130 Thigh (Experimental): Single low dose of BI 655130 administered as one single subcutaneous injection (given as 1 x 2 milliliter (mL)) in the thigh region following an overnight fast of at least 10 hours.
  Interventions: Drug: T2 - Low dose of BI 655130
- T3 - High dose of BI 655130 Periumbilical (left and right) (Experimental): Single high dose of BI 655130 administered as two single subcutaneous injections (given as 2 x 2 milliliter (mL)) in the periumbilical region (left and right) following an overnight fast of at least 10 hours.
  Interventions: Drug: T3 - High dose of BI 655130

INTERVENTIONS:
Drug: R - Low dose of BI 655130 — Single low dose of BI 655130 administered as one single subcutaneous injection (given as 1 x 2 milliliter (mL)) in the periumbilical region following an overnight fast of at least 10 hours.
  Arms: R - Low dose of BI 655130 Periumbilical
Drug: T1 - Low dose of BI 655130 — Single low dose of BI 655130 administered as two single subcutaneous injections (given as 2 x 1 milliliter (mL)) in the periumbilical region (left and right) following an overnight fast of at least 10 hours.
  Arms: T1 - Low dose of BI 655130 Periumbilical (left and right)
Drug: T2 - Low dose of BI 655130 — Single low dose of BI 655130 administered as one single subcutaneous injection (given as 1 x 2 milliliter (mL)) in the thigh region following an overnight fast of at least 10 hours.
  Arms: T2 - Low dose of BI 655130 Thigh
Drug: T3 - High dose of BI 655130 — Single high dose of BI 655130 administered as two single subcutaneous injections (given as 2 x 2 milliliter (mL)) in the periumbilical region (left and right) following an overnight fast of at least 10 hours.
  Arms: T3 - High dose of BI 655130 Periumbilical (left and right)

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of BI 655130 administered as two subcutaneous injections in the left and right periumbilical region compared to a single subcutaneous periumbilical injection of BI 655130.

The secondary objective is to investigate the relative bioavailability of a single subcutaneous injection of BI 655130 into the thigh compared to a single subcutaneous periumbilical injection of BI 655130.

ELIGIBILITY:
Inclusion Criteria:- Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests

* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 19.0 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom:

    ---implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 IU/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication up to 4 weeks after administration
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Female subjects will not be allowed to participate if any of the following applies:

* Positive pregnancy test, pregnancy or plans to become pregnant up to study completion
* Lactation

In addition, the following trial-specific exclusion criterion applies:

- Previous use of the trial medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Thoma C, Haeufel T, Li X. Assessment of the Pharmacokinetics and Safety of Spesolimab, a Humanised Anti-interleukin-36 Receptor Monoclonal Antibody, in Healthy Non-Japanese and Japanese Subjects: Results from Phase I Clinical Studies. Clin Pharmacokinet. 2022 Dec;61(12):1771-1787. doi: 10.1007/s40262-022-01176-5. Epub 2022 Dec 1. PMID 36451029
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single dose, mono-centric, open-label study in matched-group design, that is, subjects assigned to the 3 test treatment groups were matched on an individual level for gender and body weight to subjects assigned to the reference treatment group.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh | T3 - High Dose of BI 655130 Periumbilical (Left and Right)
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who received at least one dose of study drug. This was the full analysis set population in the sense of ICH-E9. It was used for analysis of safety, demographic data, and baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh | T3 - High Dose of BI 655130 Periumbilical (Left and Right) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.5) | 37.1 (5.7) | 37.4 (7.5) | 35.2 (9.2) | 35.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 10 | 40
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 12 | 12 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 11 | 11 | 12 | 12 | 46
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). Participants assigned to the Test Treatment Groups T1 and T2 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
Time Frame: Within 3 hours (h) before and 2, 3, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856, 3528 and 4200 hours following administration of the trial drug.
Population: Pharmacokinetic (PK) parameter set: all participants in the Treated set (all participants who received at least one dose of study drug) who provided at least one primary or secondary PK parameter that was not excluded because of important protocol deviations relevant to the statistical evaluation of PK endpoints or because of non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: day * microgram / milliliter
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh
Number analyzed (Participants) | 12 | 12 | 12
day * microgram / milliliter | 1227.91 (NA) — The Standard Error is geometric standard error = 1.08. | 1150.18 (NA) — The Standard Error is geometric standard error = 1.08. | 1718.47 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T1 - Low Dose of BI 655130 Periumbilical (Left and Right); Exploratory trial, no formal hypotheses were tested. Analysis of Variance (ANOVA) model on the logarithmic scale was used which included effects accounting for sources of variation: 'treatment' (fixed effect), 'matched pair' (random effect). For each matched pair in the study (participant in test treatment group matched to participant in reference treatment group), a pair number was assigned for analysis purpose; Test type: Other — Relative bioavailability; Ratio of the geometric means (T1/R) [%] = 93.67, 90% CI 2-sided [78.48 to 111.80] — The geometric means are adjusted by treatment. The geometric Coefficient of (within matched pair) Variation (gCV) [%] = 26.0
Statistical Analysis 2: Comparison: R - Low Dose of BI 655130 Periumbilical vs T2 - Low Dose of BI 655130 Thigh; [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T2/R) [%] = 139.95, 90% CI 2-sided [117.26 to 167.03] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz), Dose-Normalized
Description: Area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz), dose-normalized. Participants assigned to the Test Treatment Group T3 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
  mL = milliliter, mg = milligram.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: day * microgram * (1 / mL) * (1 / mg)
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T3 - High Dose of BI 655130 Periumbilical (Left and Right)
Number analyzed (Participants) | 12 | 12
day * microgram * (1 / mL) * (1 / mg) | 4.09 (NA) — The Standard Error is geometric standard error = 1.08. | 4.99 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T3 - High Dose of BI 655130 Periumbilical (Left and Right); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T3/R) [%] = 121.84, 90% CI 2-sided [102.08 to 145.41] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Measured Concentration of BI 655130 in Plasma (Cmax)
Description: Maximum measured concentration of BI 655130 in plasma (Cmax). Participants assigned to the Test Treatment Groups T1 and T2 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: microgram / milliliter
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh
Number analyzed (Participants) | 12 | 12 | 12
microgram / milliliter | 24.56 (NA) — The Standard Error is geometric standard error = 1.08. | 24.35 (NA) — The Standard Error is geometric standard error = 1.08. | 38.36 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T1 - Low Dose of BI 655130 Periumbilical (Left and Right); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T1/R) [%] = 99.17, 90% CI 2-sided [83.77 to 117.39] — The geometric means are adjusted by treatment. The geometric Coefficient of (within matched pair) Variation (gCV) [%] = 24.8
Statistical Analysis 2: Comparison: R - Low Dose of BI 655130 Periumbilical vs T2 - Low Dose of BI 655130 Thigh; [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T2/R) [%] = 156.20, 90% CI 2-sided [131.95 to 184.90] — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: Maximum Measured Concentration of BI 655130 in Plasma (Cmax), Dose-Normalized
Description: Maximum measured concentration of BI 655130 in plasma (Cmax), dose-normalized. Participants assigned to the Test Treatment Group T3 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: (microgram / milliliter) / milligram
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T3 - High Dose of BI 655130 Periumbilical (Left and Right)
Number analyzed (Participants) | 12 | 12
(microgram / milliliter) / milligram | 0.08 (NA) — The Standard Error is geometric standard error = 1.08. | 0.11 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T3 - High Dose of BI 655130 Periumbilical (Left and Right); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T3/R) [%] = 138.34, 90% CI 2-sided [116.87 to 163.77] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞). Participants assigned to the Test Treatment Groups T1 and T2 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: day * microgram / milliliter
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh
Number analyzed (Participants) | 12 | 12 | 12
day * microgram / milliliter | 1243.29 (NA) — The Standard Error is geometric standard error = 1.08. | 1163.47 (NA) — The Standard Error is geometric standard error = 1.08. | 1737.28 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T1 - Low Dose of BI 655130 Periumbilical (Left and Right); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T1/R) [%] = 93.58, 90% CI 2-sided [78.11 to 112.11] — The geometric means are adjusted by treatment. The geometric Coefficient of (within matched pair) Variation (gCV) [%] = 26.6
Statistical Analysis 2: Comparison: R - Low Dose of BI 655130 Periumbilical vs T2 - Low Dose of BI 655130 Thigh; [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T2/R) [%] = 139.73, 90% CI 2-sided [116.64 to 167.40] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞), Dose-Normalized
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞), dose-normalized. Participants assigned to the Test Treatment Group T3 were matched for gender and body weight (±10%) to participants assigned to Reference Treatment Group R.
  mL = milliliter, mg = milligram.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: day * microgram * (1 / mL) * (1 / mg)
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T3 - High Dose of BI 655130 Periumbilical (Left and Right)
Number analyzed (Participants) | 12 | 12
day * microgram * (1 / mL) * (1 / mg) | 4.14 (NA) — The Standard Error is geometric standard error = 1.08. | 5.03 (NA) — The Standard Error is geometric standard error = 1.08.
Statistical Analysis 1: Comparison: R - Low Dose of BI 655130 Periumbilical vs T3 - High Dose of BI 655130 Periumbilical (Left and Right); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ratio of the geometric means (T3/R) [%] = 121.34, 90% CI 2-sided [101.28 to 145.37] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: On-treatment-period, i.e. time of administration of study drug + 1 day + residual effect period of 112 days (16 weeks), up to 113 days.
Description: All participants who received at least one dose of study drug.
Arm/Group | R - Low Dose of BI 655130 Periumbilical | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) | T3 - High Dose of BI 655130 Periumbilical (Left and Right) | T2 - Low Dose of BI 655130 Thigh
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12 | 10/12 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R - Low Dose of BI 655130 Periumbilical (N=12) | T1 - Low Dose of BI 655130 Periumbilical (Left and Right) (N=12) | T3 - High Dose of BI 655130 Periumbilical (Left and Right) (N=12) | T2 - Low Dose of BI 655130 Thigh (N=12)
Headache (Nervous system disorders) | 9 | 4 | 5 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 3 | 3 | 6 | 2
Fatigue (General disorders) | 2 | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 6 | 5 | 2 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
07 Jan 2019: Amendment 2 was implemented after Independent Ethics Committee/Competent (Regulatory) authority approval. The residual effect period was changed from 176±3 days to 16 weeks for consistency across all clinical studies with BI 655130.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT03617835/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT03617835/SAP_001.pdf